CLINICAL TRIAL: NCT06237335
Title: A Phase 1/2, Multicenter Study Evaluating the Safety, Tolerability, and Biodistribution of RCT2100 With Single-Ascending Doses in Healthy Participants and Multiple-Ascending Doses and Proof-of-Concept in Participants With Cystic Fibrosis
Brief Title: A Phase 2 Study Evaluating Safety and Tolerability of RCT2100 (CFTR mRNA) in Healthy Participants and in Participants With CF
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ReCode Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCT2100-101; 2024-512169-15 (EudraCT Number)
Record Dates: First submitted 2024-01-23; First posted 2024-02-01 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; CF; mRNA
MeSH Terms: conditions — Cystic Fibrosis | interventions — ivacaftor

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participant and investigator masking only applies to Part 1 which is randomized. For Part 2, there is no masking, and this part is Open Label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- RCT2100 (Part 1) (Experimental): RCT2100 single dose
  Interventions: Drug: RCT2100
- Placebo (Part 1) (Placebo Comparator): Placebo single dose
  Interventions: Other: Placebo
- RCT2100 (Part 2) 4 week (Experimental): RCT2100 multiple dose
  Interventions: Drug: RCT2100
- RCT2100 (Part 2) 12 week (Experimental): RCT2100 multiple dose
  Interventions: Drug: RCT2100
- Experimental: RCT2100 (Part 3) 6 week (Experimental): RCT2100 multiple dose
  Interventions: Drug: Ivacaftor; Drug: RCT2100

INTERVENTIONS:
Drug: RCT2100 — RCT2100 supplied as varying dose strengths administered via oral inhalation using nebulizer
  Arms: RCT2100 (Part 1)
Other: Placebo — Placebo of similar volumes to experimental dose strengths administered via oral inhalation using nebulizer
  Arms: Placebo (Part 1)
Drug: RCT2100 — RCT2100 supplied as varying dose strengths administered via oral inhalation using nebulizer for 4 weeks
  Arms: RCT2100 (Part 2) 4 week
Drug: RCT2100 — RCT2100 supplied at a single dose strength administered via oral inhalation using nebulizer for 12 weeks
  Arms: RCT2100 (Part 2) 12 week
Drug: Ivacaftor — ivacaftor administered orally for 6 weeks
  Arms: Experimental: RCT2100 (Part 3) 6 week
Drug: RCT2100 — RCT2100 supplied at varying dose strengths. Co- administered via oral inhalation using nebulizer for 4 weeks with ivacaftor after initial 2 weeks of ivacaftor dosing run in period
  Arms: Experimental: RCT2100 (Part 3) 6 week

SUMMARY:
This is the first-in-human study with RCT2100 and is designed to provide safety and tolerability data for future clinical studies.

DETAILED DESCRIPTION:
This is a multi-part study to assess the safety, tolerability, and biodistribution of a single ascending dose of inhaled RCT2100 administered via nebulizer to healthy participants (Part 1), the safety and tolerability of multiple-ascending doses of inhaled RCT2100 administered to participants with CF (Part 2), and the safety and tolerability of RCT2100 co-administered with ivacaftor in participants with CF (Part 3).

ELIGIBILITY:
Part 1 Major Inclusion Criteria:

* Healthy, adult, male or female, 18-55 years of age, inclusive, at screening.
* Body weight greater than or equal to 50 kg and body mass index (BMI) between 16-32 kg/m2, inclusive
* The participant has a forced expiratory volume in one second (FEV1) of at least 80% predicted
* The participant is considered by the investigator to be in good general health as determined by medical history, clinical laboratory test results, vital sign measurements, 12-lead ECG results, and physical examination findings at screening.
* Understands the study procedures in the informed consent form (ICF), and is willing and able to comply with the protocol.

Part 1 Major Exclusion Criteria:

* History or presence of clinically significant medical, surgical, clinical laboratory, or psychiatric condition or disease.
* The participant has supine blood pressure (BP) >150 mm Hg (systolic) or >90 mm Hg (diastolic), following at least 5 minutes of supine rest.
* The participant has abnormal clinical laboratory tests at screening, as assessed by the study-specific laboratory.
* The participant is a smoker or has used nicotine or nicotine-containing products 6 weeks before the first dose of study drug. Former smokers with greater than 10 pack years of smoking history are excluded.

Part 2 Major Inclusion Criteria:

* Confirmed diagnosis of CF
* Forced expiratory volume in 1 second ≥50% and ≤100% of predicted mean value for age, sex, and height
* a) Not eligible for CFTR modulators based on having mutations of CFTR gene on both alleles that are not responsive to CFTR modulator therapy OR
* b) Eligible for CFTR modulators (based on local prescribing information) but not using CFTR modulators due to intolerance or contraindications

Part 2 Major Exclusion Criteria:

* Hepatic cirrhosis with portal hypertension, moderate hepatic impairment (Child Pugh Score 7 to 9), or severe hepatic impairment (Child Pugh Score 10 to 15)
* An acute upper or lower respiratory infection, pulmonary exacerbation, or changes in therapy (including antibiotics) for sinopulmonary disease within 4 weeks before the first dose of study drug
* Lung infection with organisms associated with a more rapid decline in pulmonary status
* Arterial oxygen saturation on room air less than 94% at screening
* Treatment with a CFTR modulator (Kalydeco, Trikafta, Symdeko, Orkambi, or Alyftrek) within 12 weeks of Screening

Other protocol defined Inclusion/Exclusion criteria may apply.

Part 3 Major Inclusion Criteria:

* Confirmed diagnosis of CF
* Forced expiratory volume in 1 second ≥50% and ≤100% of predicted mean value for age, sex, and height
* a) Not eligible for CFTR modulators based on having mutations of CFTR gene on both alleles that are not responsive to CFTR modulator therapy OR
* b) Eligible for dual or triple CFTR modulators (based on local prescribing information) but not using CFTR modulators due to intolerance or contraindications

Part 3 Major Exclusion Criteria:

* Hepatic cirrhosis with portal hypertension, moderate hepatic impairment (Child Pugh Score 7 to 9), or severe hepatic impairment (Child Pugh Score 10 to 15)
* An acute upper or lower respiratory infection, pulmonary exacerbation, or changes in therapy (including antibiotics) for sinopulmonary disease within 4 weeks before the first dose of study drug
* Lung infection with organisms associated with a more rapid decline in pulmonary status
* Arterial oxygen saturation on room air less than 94% at screening
* Treatment with a CFTR modulator (Kalydeco, Trikafta, Symdeko, Orkambi, or Alyftrek) within 12 weeks of Screening

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 192 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Part 1: The number of participants with Adverse Events (AEs) and Serious Adverse Events (SAEs). | From Baseline Through Day 29
  Safety and tolerability as assessed by number of participants with Adverse Events (AEs) and Serious Adverse Events (SAEs)
Part 2: The number of participants with CF with AEs and SAEs. | From Day 1 through Safety Follow-up, Week 24
  Safety and tolerability of multiple-ascending doses of inhaled RCT2100 administered to participants with CF
Part 3: The number of participants with CF with AEs and SAEs. | From Day 1 through Safety Follow-up, Week 24
  To assess the safety and tolerability of RCT2100 co-administered with ivacaftor in participants with CF.

CONTACTS AND LOCATIONS:
Overall Officials: John Matthews, MBBS, MCRP, PhD, Study Chair — ReCode Therapeutics, Inc.
Locations (23):
- United States (13):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arizona, Tucson, Arizona
  - Stanford University, Palo Alto, California
  - UCSD, San Diego, California
  - National Jewish Health, Denver, Colorado
  - Emory University, Atlanta, Georgia
  - Boston Children's Hospital, Boston, Massachusetts
  - New York Medical College, Valhalla, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Washington, Seattle, Washington
- France (2):
  - Centre Hospitalier Régional Universitaire de Montpellier - Hôpital Arnaud de Villeneuve, Montpellier
  - Hôpital Necker Enfants Malades, Paris
- UMC Utrecht, Utrecht, Netherlands
- New Zealand Clinical Research (Part 1 Only), Auckland, New Zealand
- United Kingdom (6):
  - University Hospitals Birmingham, Birmingham
  - Royal Papworth Hospital, Cambridge
  - Leeds Teaching Hospitals, Leeds
  - King's College Hospital, London
  - Nottingham University Hospitals, Nottingham
  - University Hospital Southampton, Southampton

IPD SHARING:
Plan to Share IPD: No